CLINICAL TRIAL: NCT07208084
Title: Project SOAR Awakenings: Randomized Controlled Trial for Black American Women Diagnosed With Breast Cancer
Brief Title: Project SOAR (Speaking Our African American Realities) Awakenings for Black American Women Diagnosed With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Annette L Stanton, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BCRF-24-153
Record Dates: First submitted 2025-09-03; First posted 2025-10-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; African American women; Psychoeducational; Psychosocial; Randomized controlled trial; Online; Support
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project SOAR Comparison Group (Other): Black American women diagnosed with breast cancer in this arm will receive a care box with resources for Black American women diagnosed with breast cancer.
  Interventions: Behavioral: Project SOAR comparison group
- Project SOAR Awakenings intervention (Experimental): Four Project SOAR Awakenings sessions will be conducted electronically (Zoom) by experts in a group format (12-18 participants/group) with Black American women diagnosed with breast cancer. The Strong Black Woman concept and other culturally curated topics will be discussed as they apply to group members' experience of breast cancer. All women in the study will receive a care box with resources for Black American women diagnosed with breast cancer.
  Interventions: Behavioral: Project SOAR Awakenings arm

INTERVENTIONS:
Behavioral: Project SOAR Awakenings arm — Four Project SOAR Awakenings sessions will be conducted electronically (Zoom) by experts in a group format (12-18 participants/group) with Black American women diagnosed with breast cancer. The Strong Black Woman concept and other culturally curated topics will be discussed as they apply to group members' experience of breast cancer. All women in the study will receive a care box with resources for Black American women diagnosed with breast cancer.
  Arms: Project SOAR Awakenings intervention
Behavioral: Project SOAR comparison group — Black American women diagnosed with breast cancer in this arm will receive a care box with resources for Black American women diagnosed with breast cancer.
  Arms: Project SOAR Comparison Group

SUMMARY:
The goal of this clinical trial is to test an approach to promote well-being in Black American women diagnosed with breast cancer. The main questions it aims to answer are:

* Can the Project SOAR (Speaking Our African American Realities) Awakenings online intervention improve depressive symptoms in Black American women diagnosed with breast cancer?
* Can the Project SOAR (Speaking Our African American Realities) Awakenings intervention improve fatigue in Black American women diagnosed with breast cancer?
* Can the Project SOAR (Speaking Our African American Realities) Awakenings intervention improve well-being in Black American women diagnosed with breast cancer? Researchers will compare the Awakenings online intervention to a comparison condition, to see if women in the Awakenings group improve on depressive symptoms, fatigue, and well-being more than women in the comparison group. Women in the comparison condition will receive materials by mail to use on their own.

Participants will:

* be randomized (selected by chance) to take part in four Project SOAR Gatherings, which are small group, 90-minute to two-hour online discussions with other Black American women diagnosed with breast cancer and are designed to promote well-being OR to a comparison group. Rev. Dr.(Hon) Tammie Denyse, a 20-year breast cancer survivor and patient advocate, will lead the Gatherings, along with other experts.
* devote about eight hours for women in the Project SOAR Gatherings discussions and two hours for women in the comparison group.
* complete online questionnaires at the beginning of the study and one month and three months later.
* receive a box of resources (e.g., book, cup, blanket, journal) designed to promote well-being.

DETAILED DESCRIPTION:
Recruitment of participants for the Project SOAR Awakenings trial will be conducted via the website and other social media platforms of Carrie's TOUCH (https://carriestouch.org), a nonprofit organization located in Sacramento California for Black American women diagnosed with breast cancer. The president of Carrie's TOUCH is Rev. Dr.(Hon) Tammie Denyse, the Project SOAR (Speaking Our African American Realities) Awakenings co-Principal Investigator. Recruitment also will involve announcements and a flyer to parishioner rosters of the fifth district of African Methodist Episcopal (AME) churches, which comprises 15 states and with which Rev Dr.(Hon) Denyse is affiliated.

Announcements will direct women to an email and phone number to contact if they are interested in taking part in the Project SOAR Awakenings trial. When a potential participant expresses interest in the trial via email/phone, research staff will contact her to describe the trial, summarize elements of informed consent, confirm eligibility, answer any questions, and transmit the electronic baseline questionnaire to collect demographic data and reliable and valid measures of outcome variables (i.e., depressive symptoms, fatigue, well-being) and mediators (i.e., self-compassion, cancer-related coping through emotional expression, cancer-related avoidance-oriented coping). All elements of informed consent are described at the beginning of the electronic baseline questionnaire, and contact information is provided for research staff, principal investigators, and the Institutional Review Board. At the end of the description, participants are asked to click to proceed to the baseline questionnaire if they would like to take part in the study.

Upon the completion of the baseline questionnaires, women will be randomized 1:1 via an electronic platform to the Awakenings intervention or the enhanced treatment as usual (ETAU) condition. All participants then will be mailed resources constructed to promote caring for the self, including a book (Homecoming, 2022, Bryant), an article on the Strong Black Woman schema (Denyse … Stanton, 2023), a Project SOAR personal journal, a Project SOAR cup, a Rest Deck (Rest Is Resistance, 2022, Hersey), and a Project SOAR blanket. All participants also will be compensated $100 in a gift card (e.g., Target, Amazon) for their time at the three-month assessment point.

The date and time of the first intervention session will be emailed to participants randomized to the Project SOAR Awakenings intervention, with reminder phone calls. The four Project SOAR Awakenings sessions will be conducted electronically (Zoom) in group format (10-18 participants/group) by Rev. Dr.(Hon) Denyse and another interventionist, Dr. Thea Hairston, who also is expert in psychosocial interventions with Black American women, as assisted by a doctoral candidate research staff. Leaders and participants all will identify as Black American women. One session will be conducted each week over four weeks; each session will be approximately two hours long, for a total of eight hours. Women who miss any session will be encouraged to listen to the audio-recorded session via Zoom.

With encouragement of participants to read the article on the Strong Black Woman schema prior to the session, the first session, led by Rev. Dr.(Hon) Tammie Denyse, focuses on discussing the facets of the Strong Black Woman schema (i.e., suppress emotions related to cancer, prioritize caring for others over caring for the self, resist support from other people, present an image of strength, strive to achieve with insufficient resources) and challenging the harmful facets of the schema to promote self-compassion. The session will be based on the Gathering format used in the researchers' qualitative Project SOAR research, revised for therapeutic intent. With encouragement of participants to read two chapters of the book Homecoming prior to the session, the second session also will be led by Rev. Dr.(Hon) Tammie Denyse. The session will offer foundational psychoeducation and interactional exercises on managing traumatic and stressful experiences, drawing from the book Homecoming (Bryant, 2023). The third session will be led by Dr. Thea Hairston (beloveholistic.com). Dr. Hairston employs mindful movement exercises to promote self-compassion in Black American women. Conducted by Rev. Dr.(Hon) Denyse, the fourth session will summarize and reinforce the themes of prior sessions, including making an action plan for continuing to challenge the facets of the Strong Black Woman schema and enacting self-compassion.

Intervention sessions will be audio-recorded so that participants who miss sessions can listen to them via a password-protected link; the audio-recordings will be destroyed once the study is complete. There will be no paper study materials.

Immediately after the fourth session (and at the same time for ETAU participants), participants will be sent a link to complete measures of mediators and outcomes, with reminder emails/calls as needed to promote complete data collection. Measures again will be administered electronically three months after the final intervention session, with reminder emails/calls as needed. It is estimated that each of the three assessments will require no more than 45 minutes to complete, for a potential total of 135 minutes.

All data will be collected electronically over a secure platform. To minimize risks to confidentiality, all collected data will be coded by participant number. The key to this code will be kept in a password-protected and encrypted file on a HIPAA-compliant Box account hosted by UCLA, separate from all questionnaire data. The key will be accessible only to key study personnel, and no identifying information will be shared with researchers not directly involved in the study. At the end of the study, the key will be destroyed.

Collection of names and addresses of participants is necessary in order to send the study resources (e.g., books, journal) by mail. The electronic file containing names and addresses and linking those to participant numbers will be stored separately from the rest of the data, to be accessed only by study personnel.

ELIGIBILITY:
Inclusion Criteria:

* identifying as a woman at least 18 years of age (not limited to cisgender Black American women);
* identifying as Black (African) American;
* diagnosed with breast cancer of any stage and any diagnosis duration;
* able to speak and read English;
* residing in the United States;
* access to the internet/Zoom.

Exclusion Criteria:

* men diagnosed with breast cancer,
* non-English speaker
* nonresident of the United States
* no internet access

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 90 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms - Center for Epidemiologic Studies-Depression scale | Baseline, 1 month post-baseline, 4 months post-baseline
  Validated self-report measure of depressive symptoms; range = 0-60; higher scores = greater depressive symptoms
Fatigue - PROMIS Fatigue Short Form 7a; range = 7 - 35; higher scores indicate higher fatigue | Baseline, 1 month post-baseline, 4 months post-baseline
  A validated self-report measure of fatigue

SECONDARY OUTCOMES:
Well-being-World Health Organization-Five Well-Being Index; range = 0 - 25; high scores indicate higher well-being | Baseline, 1 month post-baseline, 4 months post-baseline
  A validated self-report measure of well-being

OTHER OUTCOMES:
Self-compassion - Neff Self-Kindness subscale; range = 5 - 25; higher scores indicate higher self-kindness | Baseline, 1 month post-baseline, 4 months post-baseline
  Validated self-report measure of self-compassion
Cancer-related coping through emotional expression - Emotional Approach Coping Emotional Expression subscale; range mean = 1 - 4; higher scores indicate higher coping with cancer through emotional expression; | Baseline, 1 month post-baseline, 4 months post-baseline
  Validated measure of cancer-related coping through emotional expression
Cancer-related coping through avoidance - COPE Avoidance-oriented coping subscales; range mean = 1-4; higher scores indicate higher coping with cancer through avoidance | Baseline, 1 month post-baseline, 4 months post-baseline
  Validated self-report measure of cancer-related coping through avoidance
Giscombe Superwoman Schema Questionnaire - range mean = 0 - 3; higher scores indicate greater endorsement of schema | Baseline, 4 months post-baseline
  Validated measure of the Strong Black Woman Schema
Personal legacy of strong Black women - range mean = 1 - 5; higher scores indicate greater personal legacy of strong Black women | Baseline, 1 month post-baseline, 4 months post-baseline
  Self-report measure of personal legacy of strong Black women

CONTACTS AND LOCATIONS:
Overall Officials: Annette L Stanton, PhD, Principal Investigator — University of California, Los Angeles; Tammie Denyse, MDiv Dr(Hon), Principal Investigator — Carrie's TOUCH
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared once the trial is complete and major publications have been accepted.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Anticipated 2026-2030.
Access Criteria: To be determined.

REFERENCES:
- [Background] Owoyemi P, Denyse T, Pageot YK, Martin KJ, DeLuz KD, Kim JHJ, Stanton AL. "You [God] Gotta Go Through It With Me": Black Women Navigating Spirituality During the Breast Cancer Journey. Psychooncology. 2025 Jan;34(1):e70085. doi: 10.1002/pon.70085. PMID 39853607
- [Background] Denyse T, Martin KJ, Kim JHJ, Pageot YK, Owoyemi P, DeLuz KD, Stanton AL. "No Complaining, No Crying": A Qualitative Study of the Strong Black Woman Schema in the Breast Cancer Context. Ann Behav Med. 2023 Aug 21;57(9):733-742. doi: 10.1093/abm/kaad029. PMID 37318273
- [Background] Martin KJ, Denyse T, Pageot YK, Kim JHJ, Owoyemi P, DeLuz KD, Stanton AL. "I'm Fighting for My Life": Exploring Interactions Between Black Women with Breast Cancer and Healthcare Providers. Qual Health Res. 2023 Jul;33(8-9):753-764. doi: 10.1177/10497323231168581. Epub 2023 May 22. PMID 37212719
- [Background] Denyse T, Martin KJ, Stanton AL. The Ubuntu Approach in Project SOAR (Speaking Our African American Realities): Building a robust community-academic partnership and culturally curated focus groups. Soc Sci Med. 2022 Dec;314:115452. doi: 10.1016/j.socscimed.2022.115452. Epub 2022 Oct 12. PMID 36274454